CLINICAL TRIAL: NCT06809959
Title: Bifocal Transcranial Alternating Current Stimulation Targeting the Frontoparietal Network in Stroke Patients to Enhance Network Connectivity
Brief Title: Bifocal Transcranial Alternating Current Stimulation Targeting the Frontoparietal Network in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Technical University of Twente (Other)
Responsible Party: Principal Investigator, Fanny Quandt, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: biTACS
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Hand Functions; Cerebrovascular Disease; Brain Diseases
Keywords: Stroke; Hand motor impairment; transcranial alternating current stimulation; non-invasive brain stimulation; reach-to-grasp; functional connectivity; frontoparietal network; beta oscillations; kinematic; eeg
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Brain Diseases

STUDY DESIGN:
Intervention Model Description: Participants will receive all three types of stimulation-(i) in-phase tACS, (ii) out-of-phase tACS, and (iii) sham stimulation-on separate days in a randomized order. Each session will be separated by a one-week washout period to prevent carryover effects.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-phase-tACS (Active Comparator): Patients will perform a reach-to-grasp task with their affected hand during bifocal tACS targeting the aIPS and PMv of the lesioned hemisphere during three seperat sessions. The sequence of stimulation types will be randomized.
  Interventions: Device: In-phase-tACS
- Out-of-phase-tACS (Active Comparator): Patients will perform a reach-to-grasp task with their affected hand during bifocal tACS targeting the aIPS and PMv of the lesioned hemisphere during three seperat sessions. The sequence of stimulation types will be randomized.
  Interventions: Device: Out-of-phase-tACS
- Sham -tACS (Sham Comparator): Patients will perform a reach-to-grasp task with their affected hand during bifocal tACS targeting the aIPS and PMv of the lesioned hemisphere during three seperat sessions. The sequence of stimulation types will be randomized.
  Interventions: Device: Sham -tACS

INTERVENTIONS:
Device: In-phase-tACS — 21 minutes and 30 seconds of bifocal stimulation at 3 mA peak-to-peak per field, targeting the aIPS and PMv of the lesioned hemisphere. The stimulation is delivered at 24 Hz with the waveforms of both fields aligned in phase. A 10-second ramp-up at the beginning and a 10-second ramp-down at the end are included to ensure participant comfort. The protocol is administered using the Starstim® device with gel-based electrodes, each with a π cm² surface area.
  Arms: In-phase-tACS
Device: Out-of-phase-tACS — 21 minutes and 30 seconds of bifocal stimulation at 3 mA peak-to-peak per field over the aIPS and PMv of the lesioned hemisphere at 24 Hz. In this condition, the waveforms of the two fields are shifted by 180°, creating an out-of-phase stimulation pattern. A 10-second ramp-up and ramp-down are included, and the protocol is administered using the Starstim® device with gel-based electrodes, each with a π cm² surface area.
  Arms: Out-of-phase-tACS
Device: Sham -tACS — 21 minutes and 30 seconds of stimulation mimicking the setup of active tACS, with an initial 10-second ramp-up followed by a 10-second ramp-down. The remainder of the session is stimulation-free. This protocol is administered using the Starstim® device and gel-based electrodes with a π cm² surface area, maintaining the same setup as the active conditions to ensure comparability.
  Arms: Sham -tACS

SUMMARY:
Hand and arm function is often significantly impaired in stroke patients, making its recovery a primary goal in rehabilitative treatment. This study investigates the effects of bifocal transcranial alternating current stimulation (tACS) on the frontoparietal network in stroke patients during the subacute to chronic recovery phase. By using non-invasive brain stimulation, the study aims to modulate the neural network connectivity between the ipsilesional parietal and premotor cortices. Electroencephalography and kinematic data will be utilized to assess the impact of tACS on functional connectivity and its subsequent effect on motor function. The ultimate goal is to enhance functional coupling within these networks to promote motor function in stroke patients.

DETAILED DESCRIPTION:
Hand and arm function is often significantly impaired in stroke patients, making recovery of these functions a primary goal in stroke rehabilitation. Despite advances in acute stroke thera-pies, more than 50% of stroke survivors continue to experience motor deficits, particularly in hand and arm function, which negatively impacts their quality of life. The integrity of neural networks, especially the frontoparietal network, plays a central role in motor control, and has been shown to be altered after stroke. Transcranial alternating current stimulation (tACS) offers a promis-ing approach to modulate these brain network connections, potentially influencing motor func-tion in stroke patients.

In a randomized, controlled, triple-blind, crossover design, this study investigates the effects of 24Hz bifocal tACS on functional connectivity between the ipsilesional anterior intraparietal sulcus (aIPS) and ventral premotor cortex (PMv) in stroke patients during the subacute to chronic recovery phase. Each patient will receive three types of stimulation-(i) in-phase tACS, (ii) out-of-phase tACS, and (iii) sham stimulation-in a randomized order, with a one-week washout pe-riod between sessions to avoid carryover effects. During in-phase tACS, 24Hz stimulation over aIPS and PMv will be in phase; during out-of-phase stimulation, the phase across sights will vary by 180 degrees.

Bifocal tACS will be delivered using two four-electrode montages centered over the aIPS and PMv of the lesioned hemisphere for approximately 21 minutes per session. During each session, patients will perform a Reach-to-Grasp (RTG) task three times: before stimulation, during stimu-lation, and after stimulation. Patients will perform both a pinch grip and a whole-hand grasp during the RTG task. EEG data will be collected pre- and post-stimulation, while kinematic meas-urements will also be recorded during the stimulation task. To minimize skin sensations under the electrodes and improve blinding, a local anesthetic consisting of lidocaine and prilocaine will be applied prior to electrode placement. Clinical assessments as well as structural and func-tional imaging will be obtained to characterize each patient.

The investigators hypothesize that 24Hz bifocal tACS on the frontoparietal network alters its connectivity compared to sham stimulation.

This study seeks to enhance the understanding of functional coupling within the frontoparietal network, aiming to establish bifocal tACS as a targeted and innovative therapy to improve motor function in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* First-ever clinical stroke
* Signed informed consent
* First-ever clinical ischemic stroke at least 3 months ago
* Stimulation areas (PMv and IPS) are unaffected
* Residual deficits in the upper limb

Exclusion Criteria:

* Presence of additional neurological or psychiatric disorders
* Use of psychotropic medication
* Pregnancy or potential pregnancy in female participants
* Pacemakers, other stimulators, or medication pumps
* Claustrophobia
* Non-MRI-compatible metallic implants or foreign objects in the body
* Contraindications for transcranial alternating current stimulation (e.g., epilepsy, history of seizures, any type of pacemaker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Connectivity in the frontoparietal network | Prior and after stimulation, each recording lasting 21 minutes and 30 seconds.
  Changes in beta-band functional connectivity between aIPS and PMv during the reach-to -grasp task obtained from EEG recording prior and after each session will be evaluated, and compared across stimulation types (in-phase, out-of-phase, and sham).

SECONDARY OUTCOMES:
Motor Task Performance | Three 21-minute-and-30-second measurements (before, during, and after tACS) will be conducted across three sessions for each tACS condition (in-phase, out-of-phase, and sham) with one-week intervals between sessions.
  Motor task performance will be assessed through kinematic data collected during the Reach-to-Grasp task. An exploratory kinematic analysis will investigate whether tACS stimulation enhances motor task performance compared to sham stimulation. These effects will be analyzed both within sessions and across stimulation conditions (in-phase, out-of-phase, and sham) to identify stimulation-specific influences on motor performance.
Beta power in the frontoparietal network | Prior and after stimulation, each recording lasting 21 minutes and 30 seconds.
  Changes in beta-band power over aIPS and PMv during the reach-to -grasp task obtained from EEG recording prior and after each session will be evaluated, and compared across stimulation types (in-phase, out-of-phase, and sham).

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Quandt, Dr. med., Principal Investigator — Deparment of Neurology, University Medical Center Hamburg-Eppendorf; Robert Schulz, PD Dr. med., Principal Investigator — Deparment of Neurology, University Medical Center Hamburg-Eppendorf
Locations (1):
- Department of Neurology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided